CLINICAL TRIAL: NCT07239050
Title: Effectiveness of Intraosseus Injection Using Extra-short Needle Combined With Infiltration in Pediatric Patients With Molar Incisor Hypomineralization (A Randomized Controlled Clinical Trial)
Brief Title: Intraosseus Injection Using Extra-short Needle Combined With Infiltration in Pediatric Patients With Molar Incisor Hypomineralization
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Alexandria University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1109-07/2025
Record Dates: First submitted 2025-11-16; First posted 2025-11-20 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-10

CONDITIONS: Molar Hypomineralization
MeSH Terms: conditions — Molar Hypomineralization

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intraosseous (Experimental)
  Interventions: Other: intraosseus anesthesia
- Conventional nerve block (Active Comparator)
  Interventions: Other: Conventional nerve block

INTERVENTIONS:
Other: intraosseus anesthesia — MIH-affected hypersensitive deeply carious FPM extending into the inner 1/3 of the dentin mandibular FPM allocated to be anesthesized using infiltration followed by intraosseus anesthesia using extra-short 31-G needle.
  Arms: Intraosseous
Other: Conventional nerve block — MIH affected hypersensitive deeply carious FPM extending into the inner 1/3 of the dentin mandibular FPM allocated to be anesthesized using long 30-G needle (IANB) and short 30-G short needle (buccal infiltration).
  Arms: Conventional nerve block

SUMMARY:
Background: Effective pain control is crucial in managing pediatric dental patients. Molar-incisor hypomineralization (MIH), marked by enamel defects and dentin hypersensitivity, often hinders effective local anesthesia. Traditional injection methods may fall short, causing discomfort and complicating treatment. Combining infiltration with intraosseous injection using an extra-short 31-G needle may offer a more effective alternative.

Purpose: To compare the effectiveness of combined infiltration and intraosseous injection with an extra-short 31-G needle versus conventional techniques in eliminating pain during

ELIGIBILITY:
Inclusion Criteria:

* Healthy children, American Society of Anesthesiologists class I, II
* Cooperative children during preoperative assessments according to the Frankl'
* Behavioral Rating Scale (scores 3 or 4)
* Patient presenting with at least one hypersensitive SCASS 2,3 [22] (Appendix III) deeply carious, MIH-affected FPM, with caries extending to the inner third of the dentin and close to the pulp, as shown in the periapical radiograph, consistent with TNI 4c classification for MIH
* Written consent of the legal guardian.

Exclusion Criteria:

* Any physical or mental disability or psychological problems.
* Immunocompromised patients.
* Hypersensitivity to local anesthetic drugs used.
* Taking analgesics or other medications that alter the child's behavior or awareness of pain 12- hours pre-operatively
* Patients requiring emergency treatment.
* FPM with preoperative signs and symptoms of clinical failure

Ages: 6 Years to 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 26 (Estimated)
Dates: Start 2025-11-28 (Estimated); Primary Completion 2026-01-20 (Estimated); Study Completion 2026-01-20 (Estimated)

PRIMARY OUTCOMES:
Change in objective pain reaction | throughout the procedure
  Pain response will be assessed using Face, Legs, Activity, Cry Consolability (FLACC) scale The scale has five criteria, each assigned a score of 0, 1 or 2 (zero means no pain and 2 means severe pain). The total score scale is scored in a range of 0-10 with 0 representing no pain
Change in subjective pain scores | throughout the procedure
  It will be done by the child using Wong-Baker Faces Pain Rating Scale that ranged from 0 to 5. zero means no pain and 5 means pain is severe

SECONDARY OUTCOMES:
Local anesthesia efficacy | throughout the procedure
  The Efficacy of local anesthesia to complete the restorative procedure successfully without pain will be evaluated by Efficacy Scale
change in child anxiety | throughout the procedure
  It will be assessed using Venham Clinical Anxiety Scale (VCAS)

CONTACTS AND LOCATIONS:
Locations (1):
- Outpatient clinics of Faculty of Dentistry, Alexandria University, Egypt, Alexandria, Azarita, Egypt